CLINICAL TRIAL: NCT05370365
Title: Four or Six Weeks of Immobilization in the Conservative Treatment of Distal Radius Fractures in Elderly Population?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4/6
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Prospective single-blinded randomised clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data from the demographic data collection and the outcome parameters will be cleaned blindly from the treatment data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 week cast (Experimental): Patients over 65 years old with a distal radius fracture will be treated conservatively with a cast for 4 weeks. Once the immobilization will be removed, the standard rehabilitation protocol of our center used in these fractures will be carried out. The usual clinical and radiological follow-up will be performed at 3, 6 and 12 months.
  Interventions: Procedure: Below elbow cast
- 6 week cast (Experimental): Patients over 65 years old with a distal radius fracture will be treated conservatively with a cast for 6 weeks. Once the immobilization will be removed, the standard rehabilitation protocol of our center used in these fractures will be carried out. The usual clinical and radiological follow-up will be performed at 3, 6 and 12 months.
  Interventions: Procedure: Below elbow cast

INTERVENTIONS:
Procedure: Below elbow cast — Patients will be stay with a below elbow cast for 4 or 6 weeks

SUMMARY:
The purpose of this study is to compare if there are differences in wrist function and pain after a distal radius fracture treated conservatively with immobilization for 4 or 6 weeks in elderly patients after six months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years with a low energy distal radius fracture
* Intra or extraarticular distal radius fracture (A2, A3, C1, C2)
* Acceptable primary reduction (dorsal inclination <10º, radial shortening <3mm, articular gap <2mm)

Exclusion criteria:

* History of ipsilateral fracture
* Bilateral fracture
* Open fracture
* Other concomitant fracture (except ulnar styloid fracture)
* Fracture AO B
* Previous surgeries in this area
* Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 3 months
  The PRWE is a 15-item questionnaire designed to measure pain and wrist disability in activities of daily living.
Patient Rated Wrist Evaluation (PRWE) | 6 months
  The PRWE is a 15-item questionnaire designed to measure pain and wrist disability in activities of daily living.
Patient Rated Wrist Evaluation (PRWE) | 1 year
  The PRWE is a 15-item questionnaire designed to measure pain and wrist disability in activities of daily living.

SECONDARY OUTCOMES:
Quick Disability of Arm and Shoulder (QuickDASH) | 3 months
  It is a questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
Quick Disability of Arm and Shoulder (QuickDASH) | 6 months
  It is a questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
Quick Disability of Arm and Shoulder (QuickDASH) | 1 year
  It is a questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
Visual Analogue Scale (VAS) | 3 months
  is a measuring instrument that tries to measure the amount of pain a patient feels, which is supposed to be a value that oscillates in a continuous between no pain and an extreme amount of pain.
Visual Analogue Scale (VAS) | 6 months
  is a measuring instrument that tries to measure the amount of pain a patient feels, which is supposed to be a value that oscillates in a continuous between no pain and an extreme amount of pain.
Visual Analogue Scale (VAS) | 1 year
  is a measuring instrument that tries to measure the amount of pain a patient feels, which is supposed to be a value that oscillates in a continuous between no pain and an extreme amount of pain.
Range Of Movement (ROM) | 3 months
  Flexion, Extension, radial and ulnar deviation
Range Of Movement (ROM) | 6 months
  Flexion, Extension, radial and ulnar deviation
Range Of Movement (ROM) | 1 year
  Flexion, Extension, radial and ulnar deviation
Complications | 1 year
  Stiffness, delayed and non-union and complex regional pain syndrome (CRPS).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sala-Pujals A, Portes Chiva A, Chillon Soria J, Valverde Vilamala D, Dominguez Font E, Pardo Pol A. Immobilization Time for Conservative Treatment of Distal Radial Fractures in Elderly Patients: A Randomized Controlled Trial. J Bone Joint Surg Am. 2025 Jun 5;107(14):1628-1635. doi: 10.2106/JBJS.24.01480. PMID 40472139